CLINICAL TRIAL: NCT05213169
Title: Randomized Controlled Trial of Apomorphine in Severe Brain-injured Patients: a Double-blind Behavioral and Neuroimaging Study
Brief Title: Apomorphine in Severe Brain-injured Patients
Acronym: APODoC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Neurologique William Lennox (Belgium) (Unknown); Hôpital Valdor - ISoSL (Belgium) (Unknown); VITHAS hospitales (Spain) (Unknown)
Responsible Party: Principal Investigator, Olivia Gosseries, Research Associate, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/81b
Record Dates: First submitted 2021-12-20; First posted 2022-01-28 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Disorder of Consciousness
Keywords: unresponsive wakefulness syndrome; minimally conscious state; apomorphine; treatment
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Apomorphine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Apomorphine treatment or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apomorphine (Experimental): Apomorphine hydrochloride subcutaneous infusion 12 hours per day during 30 days: titration phase from 0 to 4 mg/h (5 days), maintenance phase at 4 mg/h, titration-maintenance phase with possible increase up to 6 mg/h depending on tolerance (18 days).
  Domperidone 20mg t.i.d per os (or via gastric tube) will be initiated to reduce common side effects 2 days before the initiation of apomorphine and maintained at least 7 days before an optional tapering off in the absence side effects.
  Interventions: Drug: Apomorphine Hydrochloride 5mg/ml
- Isotonic saline (Placebo Comparator): Sodium chloride infusion following the administration procedure described for apomorphine
  Interventions: Other: Sodium chloride 9mg/ml

INTERVENTIONS:
Drug: Apomorphine Hydrochloride 5mg/ml — Product administered using an external continuous subcutaneous infusion pump.
  Arms: Apomorphine
Other: Sodium chloride 9mg/ml — Product administered using an external continuous subcutaneous infusion pump.
  Arms: Isotonic saline

SUMMARY:
Background:

Patients who survive severe brain injury may develop chronic disorders of consciousness (DoC). Treating these patients to improve recovery is extremely challenging because of scarce and inefficient therapeutical options. Among pharmacological treatments, apomorphine, a potent direct dopamine agonist, has exhibited promising behavioral effects, but its true efficacy and its mechanism remains unknown. This randomized controlled study aims to verify the effects of apomorphine subcutaneous infusion in patients with disorders of consciousness and investigate the neural networks targeted by this treatment.

Methods/design:

The double-blind randomized controlled trial will include 48 patients: 24 patients will be randomly assigned to the apomorphine and 24 to the placebo group. Investigators and the patients will be unaware of the nature of the treatment rendered.

Primary outcome will be determined as behavioral response to treatment as measured by changes of diagnosis using the Coma Recovery Scale - Revised (CRS-R), while secondary outcome measures will include the Nociception Coma Scale - Revised (NCS-R), Disability Rating Scale (DRS), Wessex Head Injury Matrix (WHIM), circadian rhythm using actimetry, electroencephalography (EEG), positron emission tomography (PET) and functional magnetic resonance imaging (fMRI). The Glasgow Outcome Scale - Extended (GOS-E) and a phone-adapted version of the CRS-R will be used for long-term follow-up.

Statistical analyses will focus on the detection of changes induced by apomorphine treatment at the individual level (comparing data before and after treatment) and at the group level (comparing responders with non-responders). Response to treatment will be measured at four different levels: 1. behavioral response (CRS-R, NCS-R, DRS, WHIM, GOS-E, phone CRS-R), 2. brain metabolism (PET), 3. network connectivity (resting-state fMRI, clinical EEG and high-density EEG) and 4. Circadian rhythm changes (actimetry, body temperature, 24h-EEG).

Discussion:

Apomorphine is a promising and safe strategy for the treatment of DoC but efficacy, profile of the responding population and underlying mechanism remain to be determined. This trial will provide unprecedented data that will allow to investigate the response to apomorphine using multimodal methods and shed new light on the brain networks targeted by this drug in terms of behavioral response, functional connectivity and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old.
* Clinically stable, not dependent on medical ventilators for respiration.
* Diagnosed as in an unresponsive wakefulness syndrome or minimally conscious state according to the international criteria and based on at least 2 consistent CRS-R in the last 14 days (one CRS-R in the last 7 days).
* More than 4 weeks post-insult.
* No serious neurological impairments others than related to their acquired brain injury.
* No neurological medications other than anti-epileptic or anti-spasticity drugs within the last two weeks.
* No use of dopaminergic medications other than apomorphine within the last two weeks.
* Informed consent from legal representative of the patient (if patients recover, their consent will also be obtained).

Exclusion Criteria:

* Use of dopamine agonists or antagonists (e.g. amantadine, bromocriptine, l-dopa, pramipexole, ropinirole, amphetamine, bupropion, methylphenidate / risperidone, haloperidol, chlorpromazine, flupentixol, clozapine, olanzapine, quetiapine) in the last 4 weeks or 4 half-lives of the drug.
* Use of drugs with known significant prolongation of the QT interval (e.g. class 1 antiarrythmics, sotalol, macrolides, quinolones, antipsychotic drugs, tricyclic antidepressants. Methadone, chloroquine, quinine)
* A corrected QT interval over 480ms (calculated using Bazett's formula on a standard 12-lead ECG recorded in the last 14 days) or other risk factors for arrhythmia (congestive cardiac failure, severe hepatic impairment or significant electrolyte disturbance).
* A history of previous neurological functional impairment.
* Contraindication to MRI, EEG, or PET (e.g., electronic implanted devices, active epilepsy, external ventricular drain).
* Use of nitrates or other vasodilators, central nervous system acting agents such as barbiturates, morphine and related drugs (relative exclusion criterion)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Coma Recovery Scale - Revised (CRS-R) | up to 90 days (5 CRS-R baseline, 5 CRS-R treatment, 5 CRS-R follow-up)
  The CRS-R is a standardized validated neurobehavioral scale designed to assess patients with disorders of consciousness. It is divided in 6 subscales: Auditory Function (0-4 points), Visual Function (0-5 points), Motor Function (0-6 points), Oromotor/Verbal Function (0-3 points), Communication (0-2 points), Arousal (0-3 points). The subscores are summed to calculate a total score ranging from 0 to 23 points. Higher scores indicate better functions. More importantly, it provides the patient's diagnosis (coma, UWS, MCS-, MCS+, EMCS) based on the presence of specific items in different subscales (regardless of total score). Analyses will look for changes of diagnosis, changes of total score and changes of each subscore before, during and after apomorphine treatment.

SECONDARY OUTCOMES:
Change from Baseline Nociception Coma Scale - Revised (NCS-R) | up to 90 days (5 NCS-R baseline, 5 NCS-R treatment, 5 NCS-R follow-up)
  The NCS-R is a standardized validated scale designed to assess the perception of pain in patients with disorders of consciousness unable to functionally communicate. It is divided in 3 subscales: Motor Response (0-3 points), Verbal Response (0-3 points) and Facial Expression (0-3 points). The subscores are summed to calculate a total score ranging from 0 to 9 points. Higher scores indicate a higher perception of pain. Analyses will look for changes of total score and changes of each subscore before, during and after treatment.
Change from Baseline Disability Rating Scale (DRS) | up to 90 days (5 DRS baseline, 5 DRS treatment, 5 DRS follow-up)
  The DRS is validated scale designed to assess disability including the impairment and handicap of patients. It is divided in 8 subscales: eye-opening (0-3 points), communication ability (0-4 points), motor response (0-5 points), feeding (0-3 points), toileting (0-3 points), grooming (0-3 points), level of functioning (0-5 points) and employability (0-3 points). The subscores are summed to calculate a total score ranging from 0 to 29 points. Higher scores indicate a higher disability. Analyses will look for changes of total score before, during and after treatment.
Change from Baseline Wessex Head Injury Matrix (WHIM) | up to 90 days (5 WHIM baseline, 5 WHIM treatment, 5 WHIM follow-up)
  The WHIM is validated matrix designed to assess recovery in patients with disorders of consciousness. It is composed of 62 sequential items covering communication ability, cognitive skills and social interaction. The total number of achieved items and the highest achieved item are recorded. Analyses will look for changes of the total number and the highest achieved items before, during and after treatment.
Change from Baseline Circadian rhythm | up to 90 days (constant recording from enrollment)
  Wrist actigraph recorded data on limb movements to calculate circadian rythmycity (measured in minutes) corresponding to the period of the biological temporal rhythms with oscillations around 24 hours.
functional Magnetic Resonance Imaging (fMRI) | up to 90 days (fMRI before treatment initiation and after treatment completion)
  MRI functional connectivity using a seed-voxel approach, between regions of interest (here: striatum, globus pallidus interna, thalamus and prefrontal cortex) and the time course from all other brain voxels.
Positron Emission Tomography (PET) | up to 90 days (PET before treatment initiation and after treatment completion)
  Quantification of PET signal using standardized uptake values of fluorodeoxyglucose.
Conventional Electroencephalography (cEEG) | up to 90 days (4 cEEG baseline, 5 cEEG treatment, 5 cEEG follow-up)
  EEG spectral power within fixed bands or dynamic connectivity using median spectral connectivity and graph-theoretic topology metrics (clustering coefficient, path length, modularity and participation coefficient).
24-hour Electroencephalography (24-h EEG) | up to 90 days (24-h EEG before treatment initiation and after treatment completion)
  24-h EEG recordings to calculate the number of sleep cycles during day and night as well as the duration spent in each phase of sleep.
High-Density Electroencephalography (HD-EEG) | up to 90 days (HD-EEG before treatment initiation and after treatment completion)
  Multivariate classifier giving the probabilty to have signs of consciousness based on a machine-learning approach using 120 EEG markers.
Glasgow Outcome Scale - Extended (GOS-E) | from 6 months post-treatment up to 24 months post-treatment (GOS-E at 6 months,12 months and 24 months)
  The GOS-E is a standardized validated scale designed to assess the the functional outcome of patients with disorders of consciousness. It is a single score ranging from 1 (dead) to 8 (upper good recovery). Higher scores indicate a higher functional recovery. It will be performed remotely by telephone contact with the patient or their relatives.
  Analyses will look at differences in GOS-E score between responders and non-responders to apomorphine treatment, as well as differences in time within individual patients.
Phone-adapted CRS-R | from 6 months post-treatment up to 24 months post-treatment (phone-adapted CRS-R at 6 months,12 months and 24 months)
  The phone-adapted CRS-R is a scale designed to assess remotely patients with disorders of consciousness. Unlike the CRS-R, it does not comprise subcores or a total score, but provides the clinical diagnosis of the patient (coma, UWS, MCS-, MCS+, EMCS) using the same diagnostic items as the CRS-R.
  Analyses will look at differences in Phone-adapted CRS-R diagnosis between responders and non-responders to apomorphine treatment, as well as differences in time within individual patients.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Gosseries, Ph.D., Principal Investigator — University of Liege; Steven Laureys, M.D., Ph.D., Study Director — University hospital of Liège
Locations (4):
- Belgium (3):
  - University of Liege, Liège, Liege
  - Hôpital Valdor - ISoSL, Liège, Liège
  - Centre Hospitalier Neurologique William Lennox, Ottignies-Louvain-la-Neuve
- VITHAS, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fridman EA, Calvar J, Bonetto M, Gamzu E, Krimchansky BZ, Meli F, Leiguarda RC, Zafonte R. Fast awakening from minimally conscious state with apomorphine. Brain Inj. 2009 Feb;23(2):172-7. doi: 10.1080/02699050802649662. PMID 19191097
- [Background] Fridman EA, Krimchansky BZ, Bonetto M, Galperin T, Gamzu ER, Leiguarda RC, Zafonte R. Continuous subcutaneous apomorphine for severe disorders of consciousness after traumatic brain injury. Brain Inj. 2010;24(4):636-41. doi: 10.3109/02699051003610433. PMID 20235766
- [Background] Gosseries O, Charland-Verville V, Thonnard M, Bodart O, Laureys S, Demertzi A. Amantadine, apomorphine and zolpidem in the treatment of disorders of consciousness. Curr Pharm Des. 2014;20(26):4167-84. PMID 24025057
- [Background] Sanz LRD, Lejeune N, Blandiaux S, Bonin E, Thibaut A, Stender J, Farber NM, Zafonte RD, Schiff ND, Laureys S, Gosseries O. Treating Disorders of Consciousness With Apomorphine: Protocol for a Double-Blind Randomized Controlled Trial Using Multimodal Assessments. Front Neurol. 2019 Mar 19;10:248. doi: 10.3389/fneur.2019.00248. eCollection 2019. PMID 30941094